CLINICAL TRIAL: NCT05864131
Title: Effects of Parental Holding on Pain Response in Young Children During Cystometry: a Randomized Controlled Trial
Brief Title: Effects of Parental Holding on Pain Response in Young Children During Cystometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2021-0583
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Vesico-Ureteral Reflux; Filum Terminale Lipoma
Keywords: cystometry; children; parental holding; procedural pain; pain response; pain management
MeSH Terms: conditions — Vesico-Ureteral Reflux; Pain, Procedural; Agnosia | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lying (Active Comparator)
  Interventions: Behavioral: Lying
- Holding (Experimental)
  Interventions: Behavioral: Holding

INTERVENTIONS:
Behavioral: Lying — After the urethral catheter is inserted, the participant lies on an examination table lined with paper towels and diapers.
  Arms: Lying
Behavioral: Holding — Holding is performed as a non-pharmacological intervention to relieve pain in children during cystometry. After the urethral catheter is inserted, the participant's parent sits in the chair, placing a paper towel and diaper on their lap. The researcher lifts the participant by the shoulder and puts them on their parent's lap, and the parent holds the participant in their arms.
  Arms: Holding

SUMMARY:
Cystometry is essential for diagnosis and treatment plans by identifying the causes of lower urinary tract symptoms and objectively evaluating bladder functions in diseases such as neurogenic bladder, voiding dysfunction, and vesicoureteral reflux. Children may experience pain during this invasive procedure of inserting the urethra catheter. Furthermore, infants aged ≥ 6 months may feel pain from an unfamiliar and unnatural environment as they experience stranger anxiety. This experience can have a negative physical and emotional impact on children, and uncooperative behavioral reactions caused by pain can hinder the procedure. In this regard, parental holding is known as effective non-pharmacological procedural pain management in children. Although the International Children's Continence Society has advised performing cystometry while holding the infant as an effective non-pharmacological pain management method, there is insufficient evidence to support this. So, this study aimed to analyze the effect of parental holding on reducing pain in children during cystometry.

DETAILED DESCRIPTION:
This is an experimental study in a randomized controlled pre-posttest design. During cystometry, participants in the experimental group are placed on the parents' laps and held in the parents' arms. Participants in the control group are laid down on the examination table. The behavioral (FLACC scale) and physiological (oxygen saturation and heart rate) pain responses are measured at three time points (immediately, 3 min, and 10 min after urethral catheter insertion).

ELIGIBILITY:
Inclusion Criteria:

1. The children aged 6-18 months.
2. The children who undergo cystometry for the first time.
3. The children who undergo cystometry with their parents.

Exclusion Criteria:

1. The child who is premature or has a low birth weight
2. The primary caregiver is not the participant's parent
3. The child who has unstable vital signs
4. The child is expected to have neurological or sensory impairments (e.g., spinal cord inflammation, spina bifida).

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Behavioral pain response change measured using the FLACC(Faces, Legs, Activity, Crying, and Consolability) scale between each time point (immediately, 3 min, and 10 min after urethral catheter insertion). | Change from immediately, 3 minutes, and 10 minutes after urethral catheter insertion
  Behavioral pain response refers to facial expression changes, body movements, postures, and crying on pain stimuli. This is measured using the FLACC scale developed to evaluate acute pain in children. According to the FLACC scale, pain is rated using a total of five subcategories (Faces, Legs, Activity, Crying, and Consolability) on a scale of 0-2, and the scores are summed (range 0 to 10).
Physiological pain responses change measured using oxygen saturation (%/min). Change between each time point (immediately, 3 min, and 10 min after urethral catheter insertion), automatically measured by a Pulse oximeter. | Change from immediately, 3 minutes, and 10 minutes after urethral catheter insertion
  The oxygen saturation (%/minute) is automatically measured by a Nellcor OxiMax N-560 Pulse oximeter (Nellcor Puritan Bennett LLC, USA), and a Nellcor SpO2 sensor (Nellcor Puritan Bennett LLC, USA) is attached to the participants' toes.
Physiological pain responses change measured using heart rate (beats/min) . Change between each time point (immediately, 3 min, and 10 min after urethral catheter insertion), automatically measured by a Pulse oximeter. | Change from immediately, 3 minutes, and 10 minutes after urethral catheter insertion
  The heart rate (beats/minute) is automatically measured by a Nellcor OxiMax N-560 Pulse oximeter (Nellcor Puritan Bennett LLC, USA), and a Nellcor SpO2 sensor (Nellcor Puritan Bennett LLC, USA) is attached to the participants' toes.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing and Mo-Im Kim Nursing Research Institute, Yonsei University, Seoul, South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The authors offer the data when requested for a reasonable reason.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The authors offer the data when requested for a reasonable reason.

REFERENCES:
- [Result] Bauer SB, Nijman RJ, Drzewiecki BA, Sillen U, Hoebeke P; International Children's Continence Society Standardization Subcommittee. International Children's Continence Society standardization report on urodynamic studies of the lower urinary tract in children. Neurourol Urodyn. 2015 Sep;34(7):640-7. doi: 10.1002/nau.22783. Epub 2015 May 21. PMID 25998310
- [Result] Pancekauskaite G, Jankauskaite L. Paediatric Pain Medicine: Pain Differences, Recognition and Coping Acute Procedural Pain in Paediatric Emergency Room. Medicina (Kaunas). 2018 Nov 27;54(6):94. doi: 10.3390/medicina54060094. PMID 30486427
- [Result] Yerkes EB, Cheng EY, Wiener JS, Austin JC, Tu DD, Joseph DB, Routh JC, Tanaka ST. Translating pediatric urodynamics from clinic into collaborative research: Lessons and recommendations from the UMPIRE study group. J Pediatr Urol. 2021 Oct;17(5):716-725. doi: 10.1016/j.jpurol.2021.05.004. Epub 2021 May 11. PMID 34412976
- [Result] LoBue V, Adolph KE. Fear in infancy: Lessons from snakes, spiders, heights, and strangers. Dev Psychol. 2019 Sep;55(9):1889-1907. doi: 10.1037/dev0000675. PMID 31464493
- [Result] Hatfield LA, Ely EA. Measurement of acute pain in infants: a review of behavioral and physiological variables. Biol Res Nurs. 2015 Jan;17(1):100-11. doi: 10.1177/1099800414531448. Epub 2014 May 1. PMID 25504956
- [Result] Crellin D, Harrison D, Santamaria N, Babl FE. Comparison of the Psychometric Properties of the FLACC Scale, the MBPS and the Observer Applied Visual Analogue Scale Used to Assess Procedural Pain. J Pain Res. 2021 Mar 31;14:881-892. doi: 10.2147/JPR.S267839. eCollection 2021. PMID 33833566
- [Result] Pillai Riddell RR, Racine NM, Gennis HG, Turcotte K, Uman LS, Horton RE, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Lisi DM. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2015 Dec 2;2015(12):CD006275. doi: 10.1002/14651858.CD006275.pub3. PMID 26630545